CLINICAL TRIAL: NCT03331744
Title: Clinical Characteristics of Infantile Hemangioma: a Prospective Study
Brief Title: Clinical Characteristics of Infantile Hemangioma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi Ji, Principal Investigator, West China Hospital
Other Study IDs: 2017-118
Record Dates: First submitted 2017-10-12; First posted 2017-11-06 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Hemangioma
Keywords: Infantile hemangioma; Infantile hepatic hemangioma; Ulcerated infantile hemangioma; Clinical characteristics; Demographic characteristics
MeSH Terms: conditions — Hemangioma; Hemangioma, Capillary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary purpose of this study is to identify the clinical characteristics of infantile hemangioma (IH) in our single center in China. The second objective of the study is to identify the clinical features of infantile hepatic hemangioma (IHH) and ulceration in patients with IHs.

DETAILED DESCRIPTION:
Infantile hemangioma (IH) is the most common benign tumor of infancy with an estimated prevalence of 4%-5%. IHs may be presented in any part of body including the visceral organs, but are preferentially located on the face, head and neck area. IHs exhibit a characteristic life cycle consisting of a rapid proliferating phase within the first year of life followed by a slowly involuted phase lasting for up to five years. Although most resolve over time without major sequelae, a significant subset can result in severe complications including disfiguring and ulceration, some even could impair organ functions and threaten patients' life. Risk factors of IHs have been identified including multiple gestation, low birth weight, prematurity, white race, eclampsia and placental abnormalities. However, the exact occurrence, clinical features and risk factors of IHs is still unknown in Chinese patients because of the lack of large scale of prospective studies. In addition, characteristics of ulceration of IHs and infantile hepatic hemangiomas (IHHs) are also not well documented. Therefore, it's important to perform this prospective study to determine the clinical features of Chinese patients with IHs, and this study will also make contributions to the prevents, diagnoses and treatments of IHs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤6 years old
* Diagnose of IHs
* Consent of both parents (or the person having parental authority in families)

Exclusion Criteria:

* Congenital hemangioma, kaposiform hemangioendothelioma, or other vascular anomalies
* Age>6 years
* Hemangioma has been previous treated with corticosteroids, laser, cryotherapy, or only other treatments
* Patients with an inability to participate or to follow the study treatment and assessment plan

Max Age: 6 Years | Sex: All
Age Groups: Child
Study Population: Patients with the diagnosis of IHs will be recruited from the Department of Pediatric Surgery, West China Hospital of Sichuan University.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-10-06 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Location, size, phase of growth, morphologic subtypes, complication and outcome of IHs in patients. | 2 years
  Clinical characteristics of infantile hemangioma. Phase of growth include proliferation, plateau and involution phase. Morphologic subtypes include localized, segmental, indeterminate and multifocal type.

SECONDARY OUTCOMES:
Demographic information of IH about patient gender, birth weight, race, gestational age, prenatal testing procedures, placental abnormalities, maternal complications during pregnancy, type of fertilization and delivery type are collected. | 2 years
  Demographic characteristics in patients with IH.
Demographic information of IHH about patient gender, birth weight, race, gestational age, prenatal testing procedures, placental abnormalities, maternal complications during pregnancy, type of fertilization and delivery type are collected. | 2 years
  Demographic characteristics in patients with infantile hepatic hemangioma.
Size, type of lesion (focal, multiple and diffuse), complication and outcome of infantile hepatic hemangioma. | 2 years
  Clinical characteristics of infantile hepatic hemangioma
Location, size, complication and outcome in patients with ulcerated IHs. | 2 years
  Clinical characteristics of ulcerated IHs. Phase of growth include proliferation, plateau and involution, and morphologic subtypes include localized, segmental, indeterminate and multifocal type.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ji, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang K, Qiu T, Zhou J, Gong X, Lan Y, Zhang Z, Ji Y. Comparison of Infantile Hemangiomas in Male and Female Infants: A Prospective Study. J Dermatol. 2025 Oct;52(10):1555-1560. doi: 10.1111/1346-8138.17885. Epub 2025 Jul 25. PMID 40715016
- [Derived] Zhou J, Zhang Z, Lan Y, Yang M, Qiu T, Yang K, Zhang X, Jiang X, Hou F, Shan W, Kong F, Hu F, Chen S, Ji Y. Long-Term Outcomes of Oral Propranolol for Facial Infantile Hemangioma. Plast Reconstr Surg. 2026 Jan 1;157(1):142-149. doi: 10.1097/PRS.0000000000012186. Epub 2025 May 6. PMID 40327835
- [Derived] Gong X, Yang M, Zhang Z, Qiu T, Zhou J, Shan W, Zhang X, Lan Y, Bao P, Zhou Z, Yang C, Zhang Y, Li T, Guo J, Guo J, Lu G, Kong F, Zhang Y, Chen S, Ji Y. Clinical characteristics and managements of congenital hepatic hemangioma: a cohort study of 211 cases. Hepatol Int. 2025 Jun;19(3):682-691. doi: 10.1007/s12072-024-10756-5. Epub 2024 Nov 29. PMID 39612031
- [Derived] Gong X, Qiu T, Feng L, Yang K, Dai S, Zhou J, Zhang X, Chen S, Ji Y. Maternal and Perinatal Risk Factors for Infantile Hemangioma: A Matched Case-Control Study with a Large Sample Size. Dermatol Ther (Heidelb). 2022 Jul;12(7):1659-1670. doi: 10.1007/s13555-022-00756-4. Epub 2022 Jun 25. PMID 35751738